CLINICAL TRIAL: NCT05015855
Title: Testing Two Service Models of PrEP Delivery in OBGYN Clinics
Brief Title: Testing Two Models of PrEP Delivery in OBGYN Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: New York State Psychiatric Institute (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-13268; 5P30AI124414 (NIH)
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Hiv
Keywords: HIV; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBGYN-PrEP (Placebo Comparator): OBGYN-PrEP has 4 parts: (1) prioritize PrEP; (2) train providers in PrEP and intervention; (3) identify PrEP-appropriate women through a risk screen; and (4) monitor progress and fidelity to protocol.
  Interventions: Other: OBGYN-PrEP
- NP-PC PrEP (Experimental): NP-PC PrEP incorporates the standard of care and practices in OBGYN-PrEP but enhances access to additional skilled providers, as the PrEP provider burden is shifted to a Nurse Practitioner (NP) who will use a sex-positive approach to deliver PrEP services via telemedicine
  Interventions: Other: NP-PC PrEP

INTERVENTIONS:
Other: NP-PC PrEP — All participating providers will be provided standard education around PrEP and HIV prevention, but half of the providers will be randomized to also partner with a nurse practitioner who will provide additional consultation to patients.
  Arms: NP-PC PrEP
Other: OBGYN-PrEP — OBGYN-PrEP is based on PC4PrEP (R01MH107297) that has four steps: announce the policy that PrEP counseling is the responsibility of OBGYN providers to address the "purview paradox"; train providers to manage patients on PrEP; use a screening tool to identify women appropriate for PrEP; and implementation coaching to monitor and encourage PrEP counseling
  Arms: OBGYN-PrEP

SUMMARY:
The HIV Center for Clinical and Behavioral Studies, the Albert Einstein College of Medicine and the Alliance for Positive Change will test two healthcare models that integrate PrEP into OBGYN services. Model 1 is OBGYN-PrEP with 4 parts: (1) prioritize PrEP; (2) train providers in PrEP and intervention; (3) identify PrEP-appropriate women through a risk screen; and (4) monitor progress and fidelity to protocol. Model 2 is NP-PC PrEP in which PrEP provider burden is shifted to a Nurse Practitioner (NP) who will use a sex-positive approach to deliver PrEP services via telemedicine.

DETAILED DESCRIPTION:
The Albert Einstein College of Medicine (Einstein), the HIV Center for Clinical and Behavioral Studies (HIV Center), the Montefiore Medical Center Department of Obstetrics and Gynecology (OBGYN, Implementing Partner) and the Alliance for Positive Change (Alliance, Implementing and Community Partner) will compare two healthcare models that integrate PrEP into OBGYN services. Both models are acceptable standards of care and represent evidence-based approaches to the provision of care. This study is the first example of comparing these interventions in a head-to-head, comparative-effectiveness model. Both groups will benefit from maintained access, enhanced assessment with the PrEP screening tool, and physicians will all receive an evidence-based PrEP education seminar with supporting materials and ongoing access to education and resources. MODEL 1, OBGYN-PrEP is based on PC4PrEP (R01MH107297) that has four steps: announce the policy that PrEP counseling is the responsibility of OBGYN providers to address the "purview paradox"; train providers to manage patients on PrEP; use a screening tool to identify women appropriate for PrEP; and implementation coaching to monitor and encourage PrEP counseling. The goal is that PrEP be provided by a trusted provider with whom the patient has an ongoing relationship. In MODEL 2, NP-PC PrEP, all the same provisions and practices present in Model 1 will be present however, a telehealth opportunity with a Nurse Practitioner (NP) will be provided. A skilled and PrEP-trained NP will deliver PrEP services via telemedicine visits

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age Female (biological female at birth) Ability to speak and read English or Spanish Patient at Montefiore Medical Center, Eastchester Professional Center (EPC). No gross evidence of cognitive impairment precluding consent and participation Willing to have interview digitally recorded

Exclusion Criteria:

* <18 years of age Not a female (biological female at birth)- We have excluded transgender women because their sexual and reproductive health issues and PrEP use differ from those of biological females. Does not speak English or Spanish Not a patient at Montefiore Medical Center, Eastchester Professional Center (EPC). Gross evidence of cognitive impairment precluding consent and participation Not willing to have interview digitally recorded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Uptake of PrEP | 1 year
  We will compare the patients in the NP-PC PrEP and OBGYN-PrEP arms on number of PrEP prescriptions written per 100 patients. The proportion of prescriptions written for PrEP eligible patients will be compared between the two groups (NP-PC vs OBGYN) via chi-square test.
Acceptability of intervention | 1 year
  Acceptability will be assessed through qualitative in-depth interviews (IDIs) with OBGYN providers and PCs at Alliance at the end of the interventions to identify factors that facilitate or hinder the implementation of the intervention and to assess its acceptability. We will also conduct IDIs with 10 patients in each intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Atrio, MD, MSc, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No